CLINICAL TRIAL: NCT00611910
Title: Prospective, Randomized Trial of Drug-eluting Stents vs. Bare Metal Stents for the Reduction of Restenosis in Bypass Grafts.
Brief Title: Efficacy Study of Drug-eluting and Bare Metal Stents in Bypass Graft Lesions
Acronym: ISAR-CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02707
Record Dates: First submitted 2008-01-10; First posted 2008-02-11 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Arteriosclerosis of Arterial Coronary Artery Bypass Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DES (Experimental): drug-eluting stents
  Interventions: Device: sirolimus-eluting stent; Device: paclitaxel-eluting stent; Device: biodegradable-polymer-based sirolimus-eluting stent
- BMS (Active Comparator): bare metal stents
  Interventions: Device: bare metal stents

INTERVENTIONS:
Device: sirolimus-eluting stent — due to randomization Cypher stent will be implanted
  Other Names: Cypher
  Arms: DES
Device: paclitaxel-eluting stent — due to randomization Taxus stent will be implanted
  Other Names: Taxus
  Arms: DES
Device: biodegradable-polymer-based sirolimus-eluting stent — due to randomization a rapamycin-eluting stent with biodegradable polymer will be implanted
  Other Names: ISAR-DES, Yukon PC
  Arms: DES
Device: bare metal stents — Due to randomization one bare-metal stent will be implanted. The decision about the stent type will be up to the interventionalist
  Other Names: Multilink Vision; Driver; etc.
  Arms: BMS

SUMMARY:
The aim of this study is to compare the efficacy of drug-eluting stents and bare metal stents to reduce reblockage of bypass grafts after coronary stenting

DETAILED DESCRIPTION:
A large number of studies showed that drug-eluting stents significantly reduce in-stent restenosis and the subsequent need for target vessel revascularisation compared with bare metal stents. Although this applies to the vast majority of patients, intimal hyperplasia and in-stent restenosis have not been completely eliminated and remain to occur in certain high risk subgroups. While there is a plenty of data about the efficacy of DES in complex lesions or diabetics, no randomized data exist about the efficacy of DES in coronary artery bypass graft lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% de novo stenosis located in CABG
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory

Exclusion Criteria:

* Cardiogenic shock
* Target lesion located in the native coronary vessels.
* In-stent restenosis of CABG
* Target lesion located at internal mammary artery graft or free arterial graft
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: clopidogrel, rapamycin, paclitaxel, stainless steel.
* Inability to take clopidogrel for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2007-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary end point of the study is composite of death, myocardial infarction and target lesion revascularization at one year after stent implantation | 12 months

SECONDARY OUTCOMES:
Myocardial infarction rate | 12 months
Need of target lesion revascularization (TLR), defined as any revascularization procedure involving the target lesion due to luminal re-narrowing in the presence of symptoms or objective signs of ischemia. | 12 months
All cause death | 12 months
Stent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (4):
- Germany (4):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Bad Segeberger Kliniken, Bad Segeberg
  - Deutsches Herzzentrum Muenchen, Munich
  - Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Derived] Colleran R, Kufner S, Mehilli J, Rosenbeiger C, Schupke S, Hoppmann P, Joner M, Mankerious N, Fusaro M, Cassese S, Abdel-Wahab M, Neumann FJ, Richardt G, Ibrahim T, Schunkert H, Laugwitz KL, Kastrati A, Byrne RA; ISAR-CABG Investigators. Efficacy Over Time With Drug-Eluting Stents in Saphenous Vein Graft Lesions. J Am Coll Cardiol. 2018 May 8;71(18):1973-1982. doi: 10.1016/j.jacc.2018.03.456. PMID 29724350
- [Derived] Mehilli J, Pache J, Abdel-Wahab M, Schulz S, Byrne RA, Tiroch K, Hausleiter J, Seyfarth M, Ott I, Ibrahim T, Fusaro M, Laugwitz KL, Massberg S, Neumann FJ, Richardt G, Schomig A, Kastrati A; Is Drug-Eluting-Stenting Associated with Improved Results in Coronary Artery Bypass Grafts? (ISAR-CABG) Investigators. Drug-eluting versus bare-metal stents in saphenous vein graft lesions (ISAR-CABG): a randomised controlled superiority trial. Lancet. 2011 Sep 17;378(9796):1071-8. doi: 10.1016/S0140-6736(11)61255-5. Epub 2011 Aug 26. PMID 21872918